CLINICAL TRIAL: NCT04739488
Title: The Effects of Breathing Exercises and Inhaler Training for Chronic Obstructive Pulmonary Disease Patients on the Severity of Dyspnea and Life Quality
Brief Title: Breathibg Exercises and Inhaler Trainingfor Chronic Obstructive Pulmonary Disease (COPD) Patients
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Collaborators: Assistant Professor Pınar TEKİNSOY KARTIN (Unknown)
Responsible Party: Principal Investigator, Yasemin CEYHAN, Assistant Professor Yasemin CEYHAN, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Yasemin Ceyhan
Record Dates: First submitted 2021-01-05; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: COPD; Breathlessness; Aerocele
Keywords: COPD; Inhaler training; Breathing Exercises; Dyspnea; Quality of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: quantitative and qualitative methods
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing exercise and inhaler training (Experimental): This group were given pursed lip breathing exercise and inhaler training.
  Interventions: Device: Inhaler training; Behavioral: Breathing exercises
- inhaler training (Experimental): This group were given only inhaler training
  Interventions: Device: Inhaler training

INTERVENTIONS:
Device: Inhaler training — This training was given to both intervention groups. How the patients used their inhaler medication was evaluated. The steps to use the correct inhaler medication were taught sequentially. It was applied with the patient. At the end of the training, brochures prepared by the researchers were given to the patients.
Behavioral: Breathing exercises — This training was given only to the group that received breathing exercise and inhaler training.
  Pursed lips breathing exercises were taught to the patients. Patients were asked to continue their breathing exercise for 10 minutes before using their inhaler medication.
  Thus, it was evaluated whether breathing exercises performed before using inhaler drugs provided benefit on drug effectiveness.
  Arms: Breathing exercise and inhaler training

SUMMARY:
The most common symptom of chronic obstructive pulmonary disease (COPD) is shortness of breath and causes a decrease in the patient's quality of life. The best way to relieve shortness of breath is inhaler therapy. However, it is known that patients frequently apply this treatment incorrectly. The aim of this study is to determine the effects of breathing exercises and inhaler training for COPD patients on the severity of dyspnea and life quality.

For this, two patient groups with a total of 67 people were included in the study. While one group was trained on inhaler drug use, the other group was taught breathing exercises in addition to the inhaler drug use training. Patients were asked to continue the practices they learned regularly for 4 weeks. At the end of the study, it was observed that shortness of breath decreased and the quality of life increased in both patient groups.

ELIGIBILITY:
Inclusion Criteria:

* The individuals over the age of 18,
* Who had been diagnosed with COPD for at least three months,
* Using inhalers at least twice a day,
* Misusing their drug,
* Had not previously taken breathing exercise training
* Had not participated in a rehabilitation program

Exclusion Criteria:

* Mental disorders,
* Communication disabilities,
* Heart disease that could lead to dyspnea,
* Unstable angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-12-25 (Actual)

PRIMARY OUTCOMES:
Patient Information Form | It was administered to patients in both groups when they were first included in the study.
  Consisted of 19 questions including sociodemographic and disease features of the patients
Breathing Exercise and Inhaler Application Skill Chart | It was administered to patients in breathing ezercises and inhaler training group when they were first enrolled in the study.
  Consisted of 18 items including the steps of breathing exercises and inhaler utilization to be applied to breathing exercises and inhaler group.
Inhaler Application Skill Chart | It was administered to patients in inhaler training group when they were first enrolled in the study.
  Consisted of 10 items including only the skill of applying inhaler to be applied to the both group.
  Correct steps were evaluated as 1 point and wrong steps as 0 points. It was administered to patients when they were first enrolled in the study and when they came for control four weeks later.
COPD assessment test (CAT) | It was administered to patients in both groups when they were first enrolled in the study.
  The scale developed by Jones et al. (2009) is used to measure the health status of individuals with COPD.
St. George's respiratory questionnaire (SGRQ) | It was administered to patients in both groups when they were first enrolled in the study.
  It is a quality of life questionnaire specific to patients with COPD developed by Jones and Forde (2008).
Modified medical research council (mMRC) | It was administered to patients in both groups when they were first enrolled in the study.
  It was developed by the British Medical Research Council in order to provide information about the degree of dyspnea experienced by the patient based on the patient's activity and the patient's perception of the disease. As it is a one-dimensional scale Cronbach's α coefficient could not be calculated.

SECONDARY OUTCOMES:
COPD assessment test (CAT) | It was administered to patients in both groups when they came for control four weeks later.
  The scale developed by Jones et al. (2009) is used to measure the health status of individuals with COPD.
Breathing Exercise and Inhaler Application Skill Chart | It was administered to patients in breathing ezercises and inhaler training group when they came for control four weeks later.
  Consisted of 18 items including the steps of breathing exercises and inhaler utilization to be applied to breathing exercises and inhaler group.
Inhaler Application Skill Chart | It was administered to patients in inhaler training group when they came for control four weeks later.
  Consisted of 10 items including only the skill of applying inhaler to be applied to the both group.
  Correct steps were evaluated as 1 point and wrong steps as 0 points. It was administered to patients when they were first enrolled in the study and when they came for control four weeks later.
St. George's respiratory questionnaire (SGRQ) | It was administered to patients in both groups when they came for control four weeks later.
  It is a quality of life questionnaire specific to patients with COPD developed by Jones and Forde (2008).
Modified medical research council (mMRC) | It was administered to patients in both groups when they came for control four weeks later.
  It was developed by the British Medical Research Council in order to provide information about the degree of dyspnea experienced by the patient based on the patient's activity and the patient's perception of the disease. As it is a one-dimensional scale Cronbach's α coefficient could not be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University Faculty of Health Sciences, Kırşehir, Centrum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ceyhan Y, Tekinsoy Kartin P. The effects of breathing exercises and inhaler training in patients with COPD on the severity of dyspnea and life quality: a randomized controlled trial. Trials. 2022 Aug 26;23(1):707. doi: 10.1186/s13063-022-06603-3. PMID 36028881